CLINICAL TRIAL: NCT00989378
Title: Ancillary Studies to Major Ongoing NIDDK Clinical Research Studies
Brief Title: Individual Differences in Diabetes Risk: Role of Slow WaveSleep
Status: Completed | Type: Observational
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Other Study IDs: 16026A
Record Dates: First submitted 2009-10-01; First posted 2009-10-05 (Estimated); Last update posted 2013-09-05 (Estimated); Status verified 2013-09

CONDITIONS: Sleep; Diabetes
Keywords: sleep; insulin; diabetes; determine association between sleep characteristics and diabetes risk
MeSH Terms: conditions — Diabetes Mellitus; Insulin Resistance

STUDY DESIGN:
Observational Model: Cohort
Biospecimen Retention: Samples Without DNA — serum

GROUPS / COHORTS (1):
- control: normal healthy men and women
  Interventions: Behavioral: baseline study

INTERVENTIONS:
Behavioral: baseline study — normal bedtimes

SUMMARY:
This study will examine the relationship between the amount of slow wave sleep (deep sleep) and the ability of the body to bring the blood sugar level to a normal range after receiving glucose.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers age 18-20 with a BMI < 27kg/m2 in women and < 28 kg/m2 in men with normal findings on clinical examination, routine laboratory tests and EKG
* only subjects who have regular life styles (no shift work, no travel across time zone during the previous 4 weeks)
* habitual bedtimes between 7.0-8.5 hours/night
* do not take medications will be recruited

Exclusion Criteria:

* women taking hormonal contraceptive therapy and pregnant women will be excluded
* individuals with a history of psychiatric, endocrine, cardiac or sleep disorders will be excluded
* other exclusion criteria will be: tobacco use, habitual alcohol use of more than 1 drink per day, excessive caffeine intake of more than 300 mg per day

Ages: 18 Years to 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: normal healthy men and women
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2008-11; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Amount of Slow Wave Activity determines insulin sensitivity. | 2 days

CONTACTS AND LOCATIONS:
Overall Officials: Eve Van Cauter, Ph.D., Principal Investigator — University of Chicago
Locations (1):
- University of Chicago, Chicago, Illinois, United States